CLINICAL TRIAL: NCT01693939
Title: A Single Center Prospective Evaluation of the Post-LASIK Flap Thickness of the FS200 Femtosecond Laser Flap
Brief Title: Evaluation of the Post-LASIK Flap Thickness of the FS200 Femtosecond Laser Flap
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Durrie Vision (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FT-FS200-001
Record Dates: First submitted 2012-09-21; First posted 2012-09-26 (Estimated); Last update posted 2013-01-25 (Estimated); Status verified 2013-01

CONDITIONS: Myopia
Keywords: Lasik; Myopia; Femtosecond Laser
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FS200 Femtosecond Laser (Other): The LASIK flap will be created using the FS200 Femtosecond Laser
  Interventions: Device: FS200 Femtosecond Laser

INTERVENTIONS:
Device: FS200 Femtosecond Laser

SUMMARY:
The purpose of this study is to document the programmed flap thickness to achieved flap thickness using the FS200 femtosecond laser in performing LASIK procedure. The FS200 Femtosecond laser is a precision surgical device that is used to create a flap in a FDA approved LASIK procedure.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the thickness of the corneal flap created with the FS 200 Femtosecond laser flap during the LASIK procedure using the Visante and OptiVue OCT ultrasound devices.

ELIGIBILITY:
INCLUSION CRITERIA

The following are requirements for a potential study patient's inclusion into the study:

* Male or female in good general health, 18 years of age or older at the time of the pre-operative examination
* Patient must be able to read, comprehend and willing to give HIPPA and informed consent
* Patient is planning to undergo a bilateral LASIK procedure
* Both eyes must have a manifest refractive error from -1.00 to -7.00D spherical equivalent with less than or equal to 3.00 D of refractive astigmatism as expressed in spectacle minus cylinder form
* Both eyes must have a BSCVA of 20/25 or better
* Both eyes must demonstrate refractive stability confirmed by clinical records or previous glasses. Refractive stability shall be documented by a change of less than or equal to 0.50 diopter per year (sphere and cylinder) or as documented by clinical judgment by the investigator.

EXCLUSION CRITERIA

The following are exclusion criteria for study patients in this study:

* A patient with evidence of keratoconus, corneal irregularity, or abnormal videokeratography in either eye
* A patient requiring the use of any ocular drop(s) and/or medication(s) in either eye during the study period with the exception of ocular drops and/or medications provided by the investigator
* A patient having any surgical procedure within a week preceding the scheduled LASIK surgery
* A patient with any UNCONTROLLED systemic disease (i.e., a potential patient in whom therapy for a systemic disease is not yet stabilized )
* A patient with a history of prior intraocular or corneal surgery (including cataract extraction), clinically significant ophthalmic disease or abnormality (including, but not limited to, uncontrolled clinically significant blepharitis, clinically significant recurrent corneal erosion, clinically significant dry eye syndrome, clinically significant lens opacity, evidence of clinically significant trauma (including scarring inside the visual axis), or evidence of glaucoma or propensity for narrow angle glaucoma in either eye
* A patient with a significant history or current evidence of a medical, psychological or other disorder that, in the investigator's opinion, may increase the risk associated with study participation or may interfere with the interpretation of study results
* A patient with a history of any of the following medical conditions, or any other condition that could affect wound healing: uncontrolled diabetes, collagen vascular disease, autoimmune disease, immunodeficiency diseases, ocular herpes zoster or simplex, endocrine disorders (including, but not limited to unstable thyroid disorders and diabetes), lupus, and rheumatoid arthritis
* A female patient who is pregnant, nursing, planning a pregnancy during the study, or thinks she may be pregnant at the start of the study
* Current participation or participation within 30 days prior to the start of this study in a drug or other investigational device research study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-02; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Flap Thickness | 1 Week Postoperative visit
  The flap thickness will be measured one week postoperative using the Visante OCT and the Optivue OCT devices

SECONDARY OUTCOMES:
Change in Uncorrected Visual Acuity at 1 Day, 1 Week, and 1 Month Postoperatively | Postoperatively 1 month
  Change in Uncorrected visual acuity will be measured at 1 Day, 1 week, and 1 month postoperatively

OTHER OUTCOMES:
Postoperative Satisfaction Survey over Time | Postoperatively Day 1, Week 1, Month 1
  Subject questionnaire will be administered to evaluate overall patient satisfaction postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Daniel S. Durrie, MD, Principal Investigator — Durrie Vision
Locations (1):
- Durrie Vision, Overland Park, Kansas, United States